CLINICAL TRIAL: NCT01071226
Title: CHP 834 Unrelated and Partially Matched Related Donor Peripheral Stem Cell Transplantation With The CliniMACS Device for T and B Cell Depletion
Brief Title: Peripheral Blood Stem Cell Transplantation Using the CliniMACS Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Julie-An M. Talano, Associate Professor of Pediatrics and Director of Clinical Pediatric BMT Research, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHOP 07/216
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Malignant Diseases (ie, Leukemia, MDS, Lymphoma); Non-malignant Diseases (ie, Bone Marrow Failure Syndromes)
Keywords: Malignant and non-malignant diseases; Hematopoietic stem cell transplant; Peripheral blood progenitor cell transplant; CliniMACS device; T cell depletion
MeSH Terms: conditions — Leukemia; Lymphoma; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1 (Experimental): Patients receiving an unrelated donor or partially matched related donor.
  Interventions: Device: CliniMACS (CD+3, CD+19 depletion); Other: HSCT
- Stratum 2 (Experimental): For the patient's whose donors are haploidentical or a 2 antigen mismatched where one of the mismatches includes DRB1
  Interventions: Device: CliniMACS (CD 34+ positive selection); Other: HSCT

INTERVENTIONS:
Device: CliniMACS (CD+3, CD+19 depletion) — Patient's in Stratum 1 will receive grafts that have undergone CD3+, CD19+ depletion
  Arms: Stratum 1
Device: CliniMACS (CD 34+ positive selection) — Patient's in Stratum 2 will receive peripheral blood progenitor cells that have undergone CD34+ selection
  Arms: Stratum 2
Other: HSCT — Peripheral Blood Stem Cell Transplant

SUMMARY:
T cell depletion utilizing the CliniMACS device will allow more precise, specific and controlled graft engineering of peripheral blood stem cells from unrelated and partially matched related donors without an increase in relapse or graft rejection and grade III or IV acute graft versus host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* All races are eligible
* Malignant diseases: Leukemias and Lymphomas
* Non-malignant diseases: Severe Aplastic Anemia, immunodeficiencies

Exclusion Criteria:

* Lansky or Karnofsky > 70
* Echo > 27% shortening fraction
* renal function:serum creatinine < 1.5 x for normal age
* no active untreated infection
* DLCO > 50% of predicted value
* Hepatic: AST and ALT < 3x upper limit of normal; bilirubin < 2.0.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2016-08 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
To measure the incidence and quality of engraftment | Weekly for first 100 days, 6 months and 1 year

SECONDARY OUTCOMES:
Evaluate the incidence of acute Graft versus Health Disease and treatment related mortality. | weekly for the first 100 days and then 6 and 12 months post transplant date

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Talano, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States